CLINICAL TRIAL: NCT05568420
Title: Investigation of the Potential Effects of Pharmacologic Agents on Young Onset- Colorectal Cancer
Brief Title: A Study of the Possible Effects of Medication on Young Onset Colorectal Cancer (YOCRC)
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Shaare Zedek Medical Center (Other); Technion, Israel Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 22-254
Record Dates: First submitted 2022-09-30; First posted 2022-10-05 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer
Keywords: Pharmacologic; Colectomy specimens; 22-254
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, Blood and Tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal Cancer Cohort: * Stool collection prior to starting treatment (i.e. chemotherapy, chemoradiotherapy, etc.)
  * Blood sample to be collected either prior to starting treatment (i.e. chemotherapy, chemoradiotherapy, etc.) or during surveillance.
  * Prospective tissue collection will be utilized from clinically indicated diagnostic colonoscopies/biopsies/resections s, including surveillance colonoscopies. Non-diagnostically indicated tissue collections will not be performed. Some EOCRC patients will have already undergone prior surgical resection, with tissue (including normal colonic mucosae distant from the malignant tumor). The pathology FFPE blocks may be used as a source of normal colon tissue for genomic analysis.
- Healthy Control Cohort: Tissue collection of normal colon mucosa will be utilized from clinically indicated colonoscopies or from tissue obtained from a prior colonoscopy, non-diagnostically indicated tissue collections will not be performed. Colonoscopies for indications of IBD, anemia, and/or genetic predisposition will be excluded.
  * Stool samples will be collected at time of colonoscopy. Samples to be collected either within 3-14 days before or at least 14 days after colonoscopy, to avoid changes in microbiome caused by colonoscopy prep.
  * Blood samples will be collected at time of colonoscopy.
  * Risk factor questionnaire will be completed at time of colonoscopy. Will also try to collect stool from healthy control patients; however, if accrual is low after 3-6 months, remainder of cohort will be filled with specimen data from the Human Microbiome Project Data Portal.

SUMMARY:
This study will collect biospecimens (including blood, tissue, and stool samples) and health information to create a database-a type of collection of information-for better understanding young onset colorectal cancer (YOCRC). The study will include both people with YOCRC and healthy people.

ELIGIBILITY:
Inclusion Criteria:

CRC Cohort:

* 18-49 years old
* Histological or cytological diagnosis of colorectal adenocarcinoma
* Planned CRC resection biopsy, or colonoscopy ,including surveillance colonoscopies and/or have already undergone prior surgical resection, with tissue, including normal colonic mucosae distant from the malignant tumor (only patients providing tissue sample)
* Enrollment in IRB# 20-315, Young Onset Gastrointestinal Cancer Prospective Registry (Andrea Cercek, PI)

Healthy Control Cohort:

* 18-49 years old at time of diagnosis
* Scheduled for standard-of-care colonoscopy at MSK
* Underwent surgical resection of a traumatic injury to the colon at Shaare Zedek Medical Center (SZMC)

Exclusion Criteria:

* CRC Cohort:
* Antibiotic use within 6 months of collection of stool for gut microbiome analysis s (only patients providing stool sample)
* Known inherited cancer susceptibility gene
* History of inflammatory bowel disease

Healthy Control Cohort:

* Antibiotic use within 6 months of collection of stool for gut microbiome analysis (only patients providing stool sample)
* History of or prior treatment for cancer ≤ 5 years prior to registration. Exceptions include non-melanoma skin cancer, ductal carcinoma in situ, bladder carcinoma in situ, or carcinoma-in-situ of the cervix.
* Colonoscopy for indications of IBD, anemia and/or genetic predisposition (only patients providing tissue sample).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Potential research subjects will be identified through the Center for Young Onset Colorectal and Gastrointestinal Cancer, a member of the patient's treatment team, the principal and coprincipal investigator, or research team at Memorial Sloan Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
genomic analysis of tissue | 3 years
  For the genomic analyses, we will perform whole exome sequencing, MSK-IMPACT DNA-methylation and RNA assays of normal colonic mucosa and tumor. Other genomic analysis may be performed depending on the results of the initial analysis developments in this field. We will compare normal mucosa plus tumor in YOCRC vs normal mucosa in controls (using biopsies collected during outpatient colonoscopies not associated with hospitalizations)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cercek, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm